CLINICAL TRIAL: NCT01732549
Title: A Randomised, Double-Blind, Placebo-Controlled Proof Of Concept Study Of Maintenance Therapy With Tasquinimod In Patients With Metastatic Castrate-Resistant Prostate Cancer Who Are Not Progressing After A First Line Docetaxel Based Chemotherapy
Brief Title: A Proof of Concept Study of Maintenance Therapy With Tasquinimod in Patients With Metastatic Castrate-resistant Prostate Cancer Who Are Not Progressing After a First Line Docetaxel Based Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Development of tasquinimod in prostate cancer discontinued
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8-55-58102-002; 2012-001038-32 (EudraCT Number)
Record Dates: First submitted 2012-10-24; First posted 2012-11-26 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Castrate Resistant Prostate Cancer
MeSH Terms: interventions — tasquinimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tasquinimod (Experimental): 1 capsule daily, taken orally with water and food (0.25 mg initially then dose escalated to 0.5 mg or 1 mg per day) until disease progression or toxicity or patient's willingness to stop.
  Interventions: Drug: Tasquinimod
- Placebo (Placebo Comparator): 1 capsule daily, taken orally with water and food until disease progression or toxicity or patient's willingness to stop.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tasquinimod — A patient's dose will escalate from one level to the next, once tolerability of the current dose is established. If tolerability issues arise at 0.5 or 1 mg/day, patients will have their dose reduced to 0.25 or 0.5 mg/day, respectively.
  Arms: Tasquinimod
Drug: Placebo — Placebo capsules are identical to tasquinimod capsules in appearance and excipients but exclude the active compound (tasquinimod), to be taken orally once a day with water and food
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm that tasquinimod used as maintenance therapy is active and tolerable in patients with metastatic castrate-resistant prostate cancer not progressing after a first chemotherapy with docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented prostate cancer with evidence of metastatic disease on radiological evaluation, with or without symptoms (defined according to the BPI scale, with use of analgesics or narcotics)
* Has received a first line docetaxel based chemotherapy (as a monotherapy) every 3 weeks schedule of administration with corticosteroids for a minimum of 6 cycles with a cumulative dose ≥360 mg/m2. Any combination with investigational or non investigational agent is prohibited
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Docetaxel-related adverse effects must have been resolved to NCI-CTCAE v4.03 (Common Toxicity Criteria for Adverse Effects) Grade ≤1. Chemotherapy-induced alopecia and Grade 2 peripheral neuropathy are allowed
* No progressive disease at the end of docetaxel treatment defined according to RECIST criteria, no new lesion(s) assessed by bone scan and no elevated prostate specific antigen (PSA) for the three last tests with PSA3≤PSA2≤PSA1. The time between each PSA test should be preferably at least 14 days, however, a minimum of 7 days is acceptable.

Note: PSA value can be rounded to the nearest whole number if PSA>10 ng/mL. If the PSA3 value is above the PSA2, a fourth PSA test will be performed. The PSA4 value should be below or equal to PSA2

* Last dose of docetaxel administered between 21 and 42 days before randomisation
* Chemical or surgical castration verified by levels of serum testosterone ≤50 ng/dL (1.75 nmol/L)

Exclusion Criteria:

* Has concurrent use of other anticancer agents or treatments, with the following exceptions: ongoing treatment with luteinising hormone-releasing hormone agonists or antagonists, denosumab or bisphosphonate (e.g., zoledronic acid) is permitted if started ≥4 weeks prior to Screening. Ongoing treatment should be kept at a stable dose regimen
* Has ongoing treatment with warfarin
* Had prior radiation therapy since starting docetaxel. Exceptions may be made for palliative non-myelosuppressive radiation therapy administered more than 2 weeks prior to randomisation
* Had prior strontium, samarium or radium therapy or prior treatment with tasquinimod, or any agents with antiangiogenic properties
* Has ongoing treatment with corticosteroids at >10 mg/day prednisolone equivalent
* Has prostate cancer pain that warrants the initiation of radiotherapy or chemotherapy
* Has known brain or epidural metastases. Patients with previous medullary cord compression without any neurological deficit could be included
* Has a history of other malignancies, except adequately treated non-melanoma skin cancer or other solid tumours curatively treated, without evidence of disease for >5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (58):
- Belgium (4):
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - Leuven
  - Roeselare
- Czechia (5):
  - Prague, Hradčany
  - Prague, Libeň
  - Brno
  - Olomouc
  - Prague
- Denmark (4):
  - Aalborg
  - Aarhus
  - Copenhagen
  - Herlev
- France (12):
  - Angers
  - Bordeaux
  - Clermont-Ferrand
  - Dijon
  - Lille
  - Besancon, Lyon
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot, Lyon
  - Paris
  - Saint-Herblain
  - Toulouse
  - Villejuif
- Germany (5):
  - Aachen
  - Essen
  - München
  - Nürtingen
  - Tübingen
- Hungary (3):
  - Bajcsy-Zsilinszky Kórház, Budapest
  - Országos Onkológia Intézet, Budapest
  - Uzsoki utcai Kórház, Budapest
- Italy (7):
  - Genova
  - Milan
  - Modena
  - Pavia
  - Roma
  - Rozzano
  - Torino
- Lithuania (2):
  - Kaunas
  - Vilnius
- Poland (5):
  - Gdansk
  - Gdynia
  - Olsztyn
  - Urology and Urological Oncology Department and Clinic, Wroclaw
  - Wojewódzki Szpital Specjalistyczny we Wrocławiu, Wroclaw
- Spain (6):
  - Hospital Clinic Vllarroel, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Valle de Hebrón, Barcelona
  - Elche
  - Sabadell
  - Valencia
- United Kingdom (5):
  - Leeds
  - Guy's & St Thomas NHS Foundation, London
  - The Royal Marsden NHS Trust, London
  - University College Hospitals London, London
  - Sutton

REFERENCES:
- [Derived] Fizazi K, Ulys A, Sengelov L, Moe M, Ladoire S, Thiery-Vuillemin A, Flechon A, Guida A, Bellmunt J, Climent MA, Chowdhury S, Dumez H, Matouskova M, Penel N, Liutkauskiene S, Stachurski L, Sternberg CN, Baton F, Germann N, Daugaard G. A randomized, double-blind, placebo-controlled phase II study of maintenance therapy with tasquinimod in patients with metastatic castration-resistant prostate cancer responsive to or stabilized during first-line docetaxel chemotherapy. Ann Oncol. 2017 Nov 1;28(11):2741-2746. doi: 10.1093/annonc/mdx487. PMID 29059273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed as a multicentre study at 51 investigational sites (of which 44 randomised patients) in Belgium, Czech Republic, Denmark, France, Germany, Hungary, Italy, Lithuania, Poland, Spain and United Kingdom (UK)
Pre-assignment Details: A total of 219 patients were screened and 144 patients were randomised.
Groups:
- Tasquinimod: 1 capsule daily, taken orally with water and food (0.25 mg initially then dose escalated to 0.5 mg and then to 1 mg per day) until disease progression.
  Tasquinimod: Patients received initially an oral dose of 0.25 mg/day of tasquinimod, starting on Day 1, for at least 2 weeks. Once tolerability of the 0.25 mg/day dose was established, patients received a dose increase to 0.5 mg/day for at least 2 weeks, and then increased to 1 mg/day of study treatment. Patients showing poor tolerability for the escalated doses of tasquinimod were allowed to continue study treatment at the highest individually tolerated dose
- Placebo: 1 capsule daily, taken orally with water and food until disease progression
  Placebo: Patients received Placebo capsules (identical to tasquinimod capsules) to be taken orally once a day with water and food
Period: Overall Study
Arm/Group | Tasquinimod | Placebo
Started | 71 | 73
Ongoing in Treatment Period:Data Cut-off | 12 | 12
Withdrawn During Treatment:Data Cut-off | 59 (Withdrawn during treatment period 59 (AE 13, Consent withdrawn 13, Disease progression 31, Other 2)) | 61 (Withdrawn during treatment period 61 (AE 3, Consent withdrawn 6, Disease progression 46, Other 6))
Ongoing Treatment Period:Final Analysis | 0 | 0
Withdrawn During Treatment:Final Analysi | 71 | 73
Completed | 0 | 0
Not Completed | 71 | 73
Not completed — Adverse Event | 13 | 3
Not completed — Consent withdrawn | 13 | 6
Not completed — Disease progression | 37 | 50
Not completed — Other | 8 | 14

BASELINE CHARACTERISTICS:
Population: ITT population: All randomised patients. Patients were allocated to the treatment they were randomised to. Patients randomised that have been actually dead before randomisation were not retained in the intention to treat (ITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | Tasquinimod | Placebo | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (7.18) | 69.6 (5.57) | 69.6 (6.39)
Age, Customized [Number; unit: participants]
  18 to ≤ 65 years | 18 | 17 | 35
  66 to ≤ 75 years | 40 | 45 | 85
  > 75 years | 13 | 11 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 71 | 73 | 144
Race/Ethnicity, Customized [Number; unit: participants]
  Black/African American | 0 | 1 | 1
  Caucasian/White | 52 | 58 | 110
  Multiple Race | 1 | 0 | 1
  Missing | 18 | 14 | 32
Region of Enrollment [Number; unit: participants]
  Czech Republic | 5 | 1 | 6
  Belgium | 5 | 6 | 11
  Hungary | 2 | 2 | 4
  Denmark | 6 | 13 | 19
  Poland | 4 | 3 | 7
  Italy | 9 | 5 | 14
  United Kingdom | 8 | 6 | 14
  France | 17 | 14 | 31
  Lithuania | 7 | 10 | 17
  Germany | 3 | 3 | 6
  Spain | 5 | 10 | 15
Weight [Mean (Standard Deviation); unit: kg] | 83.7 (12.57) | 83.4 (15.09) | 83.6 (13.86)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.67 (3.543) | 28.01 (4.399) | 27.84 (3.987)
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 52 | 55 | 107
  Missing | 17 | 14 | 31
ECOG Performance Status Score [Number; unit: participants] — Eastern Co-operative Oncology Group (ECOG) Score: 0=Fully active, able to carry on all pre-disease performance without restriction, 1=Restricted in physically strenuous activity, but ambulatory & able to carry out work of a light or sedentary nature, e.g. light house work, office work, 2=Ambulatory & capable of all self-care but unable to carry out any work activities. Up & about more than 50% of waking hours, 3=Capable of limited self-care,confined to bed or chair more than 50% of waking hours, 4=Completely disabled. Cannot carry on any self care. Totally confined to bed or chair, 5=Dead
  participants
    0 (Normal Activity) | 39 | 31 | 70
    1 (Restricted Activity) | 32 | 38 | 70
    Missing | 0 | 4 | 4
Region [Number; unit: participants]
  Eastern Europe | 18 | 16 | 34
  Western Europe | 53 | 57 | 110

OUTCOME MEASURES:

1. Primary Outcome: Time to Radiological Progression Free Survival [PFS]
Description: The time from the date of randomisation to the date of radiological progression or death due to any cause.
  Radiological progression was defined
  - Using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for soft tissue lesions (Eisenhauer, EJC 2009), as at least a 20% relative and a 5 mm absolute increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters recorded on study (including Screening or the appearance of one or more new lesions) for target Lesions.
  Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
  - Using Prostate Cancer Clinical Working Group in March 2008 (PCWG2) criteria for bone lesions (Scher, JCO 2008). Progression was defined as appearance of 2 or more bone lesions.
Time Frame: Every 8 weeks until disease progression documentation (approximately up to 2.5 years)
Population: Intention to treat (ITT) Population
Measure: Median (90% Confidence Interval); unit: weeks
Groups:
- Tasquinimod: 1 capsule daily, taken orally with water and food (0.25 mg initially then dose escalated to 0.5 mg and then to 1 mg per day) until disease progression.
- Placebo: 1 capsule daily, taken orally with water and food until disease progression
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 71 | 73
weeks | 31.7 [24.3 to 53.7] | 22.7 [16.1 to 25.9]
Statistical Analysis 1: Comparison: Tasquinimod vs Placebo; Stratified[a]; Test type: Superiority or Other; p = 0.0315, Log Rank — Log-rank test adjusting for presence (or absence) of visceral metastases, opioid analgesic use and region (Eastern Europe, Western Europe). Two-sided p-value
Statistical Analysis 2: Comparison: Tasquinimod vs Placebo; Unstratified[b]; Test type: Superiority or Other; p = 0.0344, Log Rank

2. Secondary Outcome: Overall Survival Based on Number of Subjects Who Died
Description: Overall survival is defined as the time from randomisation to death due to any cause.
  The number of participants who died is presented since the Median was not reached for this assessment.
  Tasquinimod: Patients censored = 63, Patients at risk (t=0) = 71 Placebo: Patients censored = 67, Patients at risk (t=0) = 73
Time Frame: Every 3 months after study treatment stop until death (approximately up to 2.5 years)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 71 | 73
participants | 8 | 6
Statistical Analysis 1: Comparison: Tasquinimod vs Placebo; Stratified[a]; Test type: Superiority or Other; p = 0.4430, Log Rank; Adjusting for presence (or absence) of visceral metastases, opioid analgesic use and region (Eastern Europe, Western Europe). One-sided p-value

3. Secondary Outcome: Time to Progression Free Survival [PFS] on Next-line Therapy (PFS 2)
Description: The time from the date of randomisation to the date of radiological progression free survival [PFS] on next-line therapy (PFS 2) or death due to any cause.
  Radiological progression was defined
  - Using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for soft tissue lesions (Eisenhauer, EJC 2009), as at least a 20% relative and a 5 mm absolute increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters recorded on study (including Screening or the appearance of one or more new lesions) for target Lesions.
  Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
  - Using Prostate Cancer Clinical Working Group in March 2008 (PCWG2) criteria for bone lesions (Scher, JCO 2008). Progression was defined as appearance of 2 or more bone lesions.
Time Frame: Every 3 months after study treatment stop (follow-up) until progression under the next line therapy (approximately up to 2.5 years)
Population: ITT Population
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 71 | 73
weeks | 19.3 [7.1 to 30.7] | 24.1 [12.6 to NA] — The data for this maximum confidence interval (CI) is not evaluable (NE), listed as Not Available (NA). Patients censored = 44 Patients at risk (t=0) = 47
Statistical Analysis 1: Comparison: Tasquinimod vs Placebo; Stratified[a]; Test type: Superiority or Other; p = 0.5219, Log Rank; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Symptomatic PFS Based on Number of Subjects Who Had Symptomatic Progression or Death
Description: Symptomatic PFS is defined as the time from the date of randomisation to the date of symptomatic progression or death due to prostate cancer, whichever occurs first [symptomatic progression as assessed by Brief Pain Inventory (BPI) and analgesic use].
  Symptomatic progression was defined by the occurrence of pain with documented disease, skeleton related adverse events.
  The median symptomatic PFS for placebo and tasquinimod groups was not reached.
  Tasquinimod: Patients censored = 48, Patients at risk (t=0) = 71 Placebo: Patients censored = 54, Patients at risk (t=0) = 73
Time Frame: Every 8 weeks until symptomatic or radiological progression documentation (approximately up to 2.5 years)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 71 | 73
participants | 23 | 19
Statistical Analysis 1: Comparison: Tasquinimod vs Placebo; Stratified[a]; Test type: Superiority or Other; p = 0.5442, Log Rank; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: Time to Further Anticancer Treatment for Prostate Cancer
Description: Time from randomisation to further treatment for prostate cancer
Time Frame: Every 3 months after study treatment stop until further anticancer therapy for prostate cancer (approximately up to 2.5 years)
Population: ITT population
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 71 | 73
weeks | 42.3 [32.0 to 58.0] | 29.0 [23.1 to 39.1]
Statistical Analysis 1: Comparison: Tasquinimod vs Placebo; Stratified[a]; Test type: Superiority or Other; p = 0.1120, Log Rank; [statistical method as in outcome 2, analysis 1]

6. Secondary Outcome: Time to Deterioration in Functional Assessment of Cancer Therapy - Prostate (FACT-P)
Description: End of Study visit (within 14 days of last dose of study treatment)
  Impact of tasquinimod on health related quality of life (QoL) - Analysis of time to deterioration in FACT-P
  The FACT-P measurement system is a validated collection of health related quality of life (HRQOL) questionnaires used to assess HRQOL in men with prostate cancer. It is appropriate for use with patients with any form of cancer and extensions of it have been used and validated in other chronic illness condition. The FACT-P is a self-administered 39-item scale comprising five domains: physical well-being, social/family well-being, functional well-being, emotional well-being and additional concerns. The individual subscale scores range from 0 to a high between 24 and 48 and the total score ranges between 0 and 156, with higher scores representing better Quality of Life (QoL)
Time Frame: Up to End of Study visit (approximately up to 2.5 years)
Population: ITT population
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 71 | 73
weeks | 8.1 [8.1 to 13.1] | 15.7 [10.6 to 16.3]
Statistical Analysis 1: Comparison: Tasquinimod vs Placebo; Stratified[a]; Test type: Superiority or Other; p = 0.2491, Log Rank; Adjusting for presence (or absence) of visceral metastases, opioid analgesic use (or not) & region (Eastern Europe, Western Europe). One-sided p-value

7. Secondary Outcome: Change From Baseline of EuroQol-5 Dimension QoL Instrument (EQ-5D) VAS Score
Description: Baseline is defined as last measurement collected prior to the first dose of study drug. End of Study visit (within 14 days of last dose of study treatment)
  The EQ-5D, a 5-item scale useful in health resource utilisation and cost comparisons between treatment groups designed for self-completion by patients consists of two pages [EQ-5 descriptive system and EQ Visual Analogue Scale(VAS)]. The EQ-5 descriptive system comprises five dimensions: mobility, self care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, severe problems. The EQ-VAS records the respondent's self-rated health on a vertical VAS. The respondents are asked to mark health status on the day of the interview on a 10cm vertical scale with end points of 0 to100. There are notes at the both ends of the scale that the bottom rate(0) corresponds to "the worst health you can imagine", and the highest rate(100) corresponds to "the best health you can imagine"
Time Frame: Baseline and End-of-study Visit (approximately up to 2.5 years)
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: Score on scale
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 39 | 50
Score on scale | -9.0 [-74 to 63] | -3.5 [-55 to 30]

8. Secondary Outcome: Safety Profile of Tasquinimod
Description: Number of subjects reporting adverse events
Time Frame: At regular intervals during the study treatment period and every 3 months during the follow-up until death (approximately up to 2.5 years)
Population: Safety Population: All patients who received at least one dose of study treatment. Patients were allocated to the treatment they actually received
Measure: Number; unit: participants
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 71 | 70
participants
  Any Treatment Emergent Adverse Event (TEAEs) | 69 | 66
  Intensity of TEAEs [Grade 3-5 (severe)] | 36 | 19
  Intensity of TEAEs [Grade 5] | 1 | 3
  Intensity of TEAEs [Grade 4] | 3 | 2
  Intensity of TEAEs [Grade 3] | 32 | 14
  Intensity of TEAEs [Grade 2 (moderate)] | 28 | 28
  Intensity of TEAEs [Grade 1 (mild)] | 5 | 19
  Causality of TEAEs [Drug Related] | 54 | 38
  Causality of TEAEs [Not Drug Related] | 15 | 28
  TEAEs Leading to Drug Withdrawal | 12 | 3
  TEAEs leading to Dose Reduction | 16 | 2
  TEAEs leading to Drug Interruption | 33 | 12
  TEAEs Leading to Death | 1 | 0
  Serious Adverse Event (SAEs) | 24 | 16
  Drug Related SAEs | 6 | 2

ADVERSE EVENTS:
Time Frame: At regular intervals during the study treatment period and every 3 months during the follow-up until death (approximately up to 2.5 years)
Description: Non-SAE details: A summary of common (incidence >5%) TEAEs is presented
Arm/Group | Tasquinimod | Placebo
Serious Adverse Events (participants affected / at risk) | 24/71 | 16/70
Other Adverse Events (participants affected / at risk) | 69/71 | 66/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tasquinimod (N=71) | Placebo (N=70)
Vomiting (Gastrointestinal disorders) | 2 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Disease progression (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Movement disorder (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 1
Biliary cyst (Hepatobiliary disorders) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tasquinimod (N=71) | Placebo (N=70)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Spinal pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Fatigue (General disorders) | 21 | 15
Asthenia (General disorders) | 17 | 10
Oedema peripheral (General disorders) | 13 | 8
Pain (General disorders) | 5 | 4
Pyrexia (General disorders) | 6 | 3
Influenza like illness (General disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 19 | 15
Constipation (Gastrointestinal disorders) | 23 | 8
Vomiting (Gastrointestinal disorders) | 9 | 9
Diarrhoea (Gastrointestinal disorders) | 9 | 6
Abdominal pain (Gastrointestinal disorders) | 9 | 4
Flatulence (Gastrointestinal disorders) | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Headache (Nervous system disorders) | 8 | 7
Paraesthesia (Nervous system disorders) | 6 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 0
Dizziness (Nervous system disorders) | 4 | 3
Cystitis (Infections and infestations) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 26 | 8
Hypertension (Vascular disorders) | 9 | 6
Onycholysis (Skin and subcutaneous tissue disorders) | 4 | 0
Weight decreased (Investigations) | 6 | 1
Insomnia (Psychiatric disorders) | 10 | 6
Depression (Psychiatric disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Urinary retention (Renal and urinary disorders) | 1 | 5
Anaemia (Blood and lymphatic system disorders) | 9 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 5

LIMITATIONS AND CAVEATS:
The study was terminated early due to the stop of the project as decided by sponsor. The trial included number of planned patients & number of events(PFS)were met to draw conclusions. Only follow-up of patients were discontinued earlier than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No